CLINICAL TRIAL: NCT04471571
Title: A Comparison of the Effectiveness of Resin Infiltration Treatment Versus a Combined Treatment of Microabrasion and Resin Infiltration for the Management of Affected Incisors in Molar Incisor Hypomineralization (MIH) Cases
Brief Title: Resin Infiltration Treatment Versus a Combined Treatment With Microabrasion for the Management of MIH Affected Incisors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Shehab, Assistant lecurer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DShehab
Record Dates: First submitted 2020-07-02; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: two-arm parallel group randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Selection bias: will be overcome by randomization and allocation concealment. Performance bias: will be overcome by standardized method of application by single operator.
  Detection bias: will be overcome by blinding of the outcome assessor. Reporting bias: All the outcomes will be reported and published.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resin infiltration group (Active Comparator): Enamel lesions for this group will be treated only by resin infiltration.
  Interventions: Other: Resin infiltration for MIH-affected incisors
- Microabrasion + resin infiltration group (Experimental): Enamel lesions for this group will be treated first by microabrasion followed by resin infiltration.
  Interventions: Other: Resin infiltration and microabrasion for MIH-affected incisors

INTERVENTIONS:
Other: Resin infiltration and microabrasion for MIH-affected incisors — MIH-affected incisors will be treated with microabrasion followed by resin infiltration as a combined treatment
  Arms: Microabrasion + resin infiltration group
Other: Resin infiltration for MIH-affected incisors — MIH-affected incisors will be treated with resin infiltration alone
  Arms: Resin infiltration group

SUMMARY:
The prevalence of molar incisor hypomineralization is relatively high. It has been reported that MIH-affected children experience a wide range of negative impacts because of having visible enamel opacities on their incisors whether these teeth show post eruptive breakdown or not. The management of MIH is challenging with a broad spectrum of treatment modalities being available. However, there are no clear guidelines available to aid in clinical decision making. Possible treatment options for anterior teeth with MIH include: Microabrasion, resin infiltration, tooth bleaching, etch-bleach and seal technique and composite restorations or veneers. It is believed that these methods could be used alone or in a combination of methods to achieve better aesthetic results.

For MIH affected-incisors microabrasion and resin infiltration are acceptable treatment options which could be used alone or in a combination. Accordingly, the aim of this study is to compare the clinical outcomes of using resin infiltration either alone or combined with microabrasion for the management of MIH affected incisors.

DETAILED DESCRIPTION:
The study will be conducted on a dental unit in postgraduate clinic of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University, Egypt.The primary hypothesis of this study is that a resin infiltration and microabrasion combined treatment will result in better clinical outcomes than using resin infiltration alone. All treatment procedures will be carried out by the principal investigator.

36 patients will be included in the study. The teeth will be randomized into two groups according to the intervention. The study involves two types of interventions:

Group 1 (resin infiltration):

The treatment will follow the manufacturer's instructions (Icon, DMG, Hamburg, Germany). The procedure involves the application of Icon-Etch, Icon-Dry as well as Icon-Infiltrant. Followed by removal of excess and then polishing of the treated surfaces.

Group 2 (Micro-abrasion followed by resin infiltration):

The Micro-abrasion agent (Opalustre, Ultradent, South Jordan, UT, USA) will be applied to the tooth for 60 seconds using a standard rubber cup attached to a low speed hand piece followed by rinsing the tooth surface with water for 20 seconds. This procedure will be repeated up to 5 times.

Resin infiltration will then be carried out as discussed before.

Vita Easyshade Advance® spectrophotometer (Vita Zahnfabrik, Sackingen, Germany) will be used to evaluate the masking color of the teeth selected in the study.

Measurements will be taken before, immediately after, 1 month, 3 months, 6 months and 12 months after treatment.

A standardized Photograph will be taken at 5 different times (before treatment, immediately afterwards, one month, 6 months and 12 months after treatment with the exact same camera and conditions. The images collected will be analyzed and evaluated by 2 different dentists.

ELIGIBILITY:
Inclusion Criteria:

1. Cooperative children aged between 7-16 years old
2. Children with MIH having enamel opacity involving at least one permanent incisor
3. MIH- affected incisors which did not receive any previous treatment
4. 1/3 of the crown should be visible in the oral cavity
5. Lesions size should be more than 1mm
6. Healthy children

Exclusion Criteria:

1. Children with systemic diseases, allergies or any dental or facial anomaly other than MIH
2. Children aged < 7 or > 16 years old
3. Uncooperative children
4. MIH patients without the affection of the incisors or with compromised incisor esthetics due to tooth surface loss, traumatic dental injury or caries
5. MIH incisors which already received any kind of treatment
6. Lesions which are smaller than 1mm in size

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in the aesthetics and amount of color masking of the lesion | 12 months
  Vita Easyshade Advance® spectrophotometer (Vita Zahnfabrik, Sackingen, Germany) will be used to evaluate the change in color of the teeth selected in the study before and after the treatment. L*, a*, and b* values will be recorded for each tooth based on the CIEL*a* b* color space. The value of color differences or color masking (∆E) will be clinically evaluated by the formula ∆E=[(∆L*)2+(∆a*)2+(∆b*). Color readings will be taken before, immediately after, 1, 3, 6, and 12 months after treatment.

SECONDARY OUTCOMES:
Change in the patient's oral health related quality of life following the treatment: Child Perceptions Questionnaire CPQ 8-10/11-14 | 12 months
  It includes evaluating the patient's Oral Health Related Quality of life (OHRQoL) before and after treatment which is measured as difference in the scores of the Child Perceptions Questionnaire CPQ 8-10/11-14 before and after treatment. There are 36 items included in the questionnaire covering four different domains: oral symptoms, function related limitations as well as emotional and social well-being. The participants should answer regarding the frequency of certain events in the last six months. There are 5 responses to choose from: 0 = Never, 1 = Once or twice, 2 = Sometimes, 3 = Often and 4 = Every day or almost every day. The total score should range from 0 to 144. Higher scores indicate low oral health related quality of life (OHRQoL).

CONTACTS AND LOCATIONS:
Overall Officials: Shehab El-Din, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almuallem Z, Busuttil-Naudi A. Molar incisor hypomineralisation (MIH) - an overview. Br Dent J. 2018 Oct 5. doi: 10.1038/sj.bdj.2018.814. Online ahead of print. PMID 30287963
- [Background] Hasmun N, Lawson J, Vettore MV, Elcock C, Zaitoun H, Rodd H. Change in Oral Health-Related Quality of Life Following Minimally Invasive Aesthetic Treatment for Children with Molar Incisor Hypomineralisation: A Prospective Study. Dent J (Basel). 2018 Nov 1;6(4):61. doi: 10.3390/dj6040061. PMID 30388743